CLINICAL TRIAL: NCT04254419
Title: Phase 1 Study of Locoregional Injections of Ex Vivo Expanded Natural Killer Cells in Children and Young Adults With Recurrent, Progressive, or Refractory Brain Tumors
Brief Title: Phase 1 Study of Locoregional Injections of Ex Vivo Expanded Natural Killer Cells
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000659
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-03

CONDITIONS: High Grade Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NK cell infusion (Experimental): The TGFβi NK cell product on this trial will be manufactured in the Cell Based Therapy (CBT) Core facility at Nationwide Children's Hospital. Donors have been identified with specific universal-donor NK cell characteristics. The NK cells are collected from these donors via apheresis and then undergo CD3 depletion followed by a 2-week expansion. TGFβi NK cells are then generated by weekly stimulation with feeder cells and cultured in IL-2 and TGFβ. After 2 weeks, the TGFβi NK cells are washed and cryopreserved for future use. The expanded donor NK cell product will be manufactured prior to subject enrollment.
  Patients will receive 3 cycles of NK cell infusions over 12 weeks. Each cycle will consist of three weekly injections followed by a rest week (week 4). If patients have stable or improved disease and additional doses are available, patients may continue to receive therapy for a total of 12 cycles.
  Interventions: Biological: NK cells

INTERVENTIONS:
Biological: NK cells — The universal donor TGFβi NK cells will be cryopreserved until they are delivered bedside for infusion. The trained staff will thaw the product by the bedside. The administration of the cells will be done via an Ommaya intra-cavitary/a programable ventriculoperitoneal (VP) shunt.
  Once the infusion is ready for administration patients will be admitted to the infusion unit for monitoring. NK cells will be administered through the Ommaya/VP shunt in approximately 3 milliliters over approximately 2-5 minutes; followed by 1.5-2 milliliter preservative-free normal saline flush over approximately 1 minute.

SUMMARY:
Each patient will receive up to 12 cycles of TGFβi NK cell infusions. Each cycle will be of 4 weeks duration. During the first 3 weeks, TGFβi NK cells will be infused once weekly. The 4th week will be a rest week. TGFβi NK cell infusions should be delivered at least 3 days apart (e.g., Friday of Week 1 and Monday of Week 2). Dose will be escalated in an inter-patient stepwise fashion consisting of 3 dose levels.

DETAILED DESCRIPTION:
A cycle is 28 days (4 weeks) consisting of weekly infusions of UD TGFβi NK cells via Ommaya or a programable ventriculoperitoneal (VP) shunt for three weeks followed by one week of rest. The dose-limiting toxicity (DLT) period is the first 28 days (4 weeks). A DLT is defined as any event that is at least possibly attributable to the TGFβi NK cell product and that occurs from the time of initial NK cell infusion through the end of the first cycle (28 days). Patients with stable or improved disease will receive up to 12 cycles of TGFβi NK cell infusions.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis:

Recurrent, refractory, or progressive malignant CNS tumor

* Patients with a histologically confirmed diagnosis of a CNS tumor that is recurrent, progressive, or refractory with the exception of diffuse midline gliomas (DMG) or Diffuse Intrinsic Pontine Gliomas (DIPG). All tumors must have histologic verification at either the time of diagnosis or recurrence.
* Patients should be deemed candidate for placement of an Ommaya reservoir placed intra-cavitary/intra-tumoral or a programable VP shunt.
* Measurable residual tumor after surgery is not required for study entry.
* Resection cavity needs to be at least 2 cm x 2 cm in two dimensions on imaging for patients deemed as candidates for an intratumoral infusion via an Ommaya reservoir.

  * Performance score: Lansky score of 50 or greater if ≤ 16 years of age or a Karnofsky score of 50 or greater if > 16 years of age. Participants who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
  * Adequate bone marrow function, without transfusion or growth factors within 21 days of NK cell administration.
  * Adequate liver function
  * Adequate Renal Function
  * Prothrombin time/international normalized ratio
  * Patients of child-bearing potential must agree to use adequate contraception
  * Adequate neurologic function defined

Prior Therapy:

* Chemotherapy

  * All patients must have received their last dose of known myelosuppressive anticancer therapy at least 21 days prior to enrollment or at least 42 days of nitrosourea.
  * For patients who have received prior bevacizumab, at least 6 weeks must have elapsed prior to enrollment.
* Biologic or investigational agent (anti-neoplastic, non-myelosuppressive):

  * Patient must have recovered from any acute toxicity potentially related to the agent and received their last dose of the investigational or biologic agent ≥ 14 days prior to study enrollment.
  * For agents with known adverse events occurring beyond 14 days after administration, this period must be extended beyond the time during which adverse events are known to occur.
  * At least 12 weeks since the completion of any immunotherapies or cell therapies.
* Radiation Therapy

  * Focal radiation therapy > 6 weeks prior to enrollment.
  * Craniospinal irradiation >12 weeks.
* Stem Cell Transplant.

Patient must be:

* ≥ 6 months since allogeneic stem cell transplant prior to enrollment with no evidence of active graft vs. host disease.
* ≥ 3 months since autologous stem cell transplant prior to enrollment.

  • Growth Factors
* Patients must be off all colony- forming growth factor(s) for at least 1 week prior to enrollment (e.g., filgrastim, sargramostim or erythropoietin).
* 2 weeks must have elapsed if patients received long-acting formulations.

  • Corticosteroids
* Patients who are receiving dexamethasone must be on a stable or decreasing dose for at least 1 week prior to enrollment.

Exclusion Criteria:

* Patients with intra- or extra-CNS metastasis or multi-focal disease.
* Patients with diffuse midline gliomas or Diffuse Intrinsic Pontine Gliomas (primary or recurrent).
* Pregnant or lactating patients.
* Participants who are receiving any other investigational agents.
* Evidence of active uncontrolled infection or unstable or severe intercurrent medical conditions.
* Any medical condition that precludes surgery.
* Patients with a known disorder that affects their immune system, such as human immunodeficiency virus (HIV), or an auto- immune disorder requiring systemic cytotoxic or immunosuppressive therapy are not eligible.
* Evidence of bleeding diathesis or use of anticoagulant medication or any medication which may increase the risk of bleeding.
* Patients who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study are not eligible.
* History or current diagnosis of any medical or psychological condition that in the Investigator's opinion, might interfere with the subject's ability to participate

Ages: 12 Months to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-03-04 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-10 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose or Recommended Phase 2 Dose (RP2D) | 36 months
  To determine the maximum tolerated dose (MTD) and/or the RP2D of UD TGFβi NK cells that have been propagated ex vivo with genetically modified feeder cells and administered using an Ommaya reservoir (into tumor cavity) or a programable ventriculoperitoneal shunt (intraventricular).
Maximum tolerated dose | 36 months
  To establish the maximum tolerated dose (MTD) of autologous natural killer cells that have been propagated ex vivo with genetically-modified feeder cells and administered intra-tumoral via Ommaya reservoir in patients with recurrent high-grade glioma. MTD will be the maximum dose at which fewer than one-third of patients experience a dose-limiting toxicity during cycle 1 of therapy

SECONDARY OUTCOMES:
Define tumor activity in children | 6 months
  To preliminarily define the antitumor activity in children with recurrent, refractory, or progressive primary malignant CNS tumors with the exception of diffuse midline gliomas and or diffuse intrinsic pontine glioma as measured by objective response rate (ORR) of UD TGFβi NK cells within the confines of a Phase I study.

OTHER OUTCOMES:
NK cell antitumor activity | 36 months
  To assess the antitumor activity based on imaging and cytology of autologous NK cell administration directly into the tumor or the resection cavity.
Assessment of the immuno-phenotype of expanded NK cells for high-grade glioma patients | 36 months
  To determine the persistence, immuno-phenotype and function of adoptively transferred expanded TGFβi NK cells and correlate the findings with the overall response.
Assessment of health-related quality-of-life of patients using patient reported outcomes measurement information system (PROMIS) | 36 months
  To assess health-related quality-of-life of patients by parent report, and when possible patient report using PROMIS.
Assessment of the immune signature based profile | 36 months
  To determine the gene expression-based immune profile of each patient's tumor (e.g., RNA-seq or NanoString).
Changes of the T-cell Receptor (TCR) Repertoires in Tumor Tissue before and after NK Cell Treatment | 36 months
  The aim is to compare the mRNA expression of specific immune genes before and after NK cell treatment. By analyzing RNA from tumor tissue, we will identify and quantify immune cells in each patient's tumor. These profiles will be linked to treatment outcomes, helping understand response or non-response. For patients whose disease progresses, the goal is to study changes in their immune cells through RNA analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Khan, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided